CLINICAL TRIAL: NCT02437357
Title: A Randomized-Controlled Trial on Metacognitive Training for Depression (D-MCT) - an New Group Intervention for Depressed Patients
Brief Title: A Trial on Metacognitive Training for Depression (D-MCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NWF-15/03
Record Dates: First submitted 2015-03-23; First posted 2015-05-07 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Depression
Keywords: Psychotherapy, Group; Metacognition; Cognitive Bias
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metacognitive Training (Experimental): D-MCT is conceptualized as a variant of cognitive behavioral therapy (CBT) that uses a metacognitive perspective to focus on the modification of cognitive biases by using creative and engaging strategies (e.g., multimedial presentation). The training seeks to enable group members to recognize and correct the often automatic and unconscious depressive thought patterns, in part by viewing this depressive thought process at a distance (i.e., depersonalizing). Besides dysfunctional assumptions about one's thought processes, more general cognitive biases, which have been identified by basic research are at the core of the D-MCT. Finally, dysfunctional coping-strategies (i.e., thought suppression, rumination as problem-solving) are discussed and modified.
  Interventions: Other: Metacognitive Training
- Positivity Training (Active Comparator): Positivity Training (PT) is a "euthymic therapy" group based on cognitive behavioral therapy (CBT) with a focus on the education and training of sensual enjoyment and pleasure. Aim of the training is to reduce depressive symptomatology by increasing the ability to enjoy and to (re-)install positive sensory experiences. Therefore, group members are informed about the impact of positive experiences on well-being and the awareness of the five senses is trained in different practical exercises (hearing, sight, smell, taste, and touch).
  Interventions: Other: Positivity Training

INTERVENTIONS:
Other: Metacognitive Training — 8 group sessions á 60 min
  Arms: Metacognitive Training
Other: Positivity Training — 8 group sessions á 60 min
  Arms: Positivity Training

SUMMARY:
The purpose of the present randomized-controlled trial is to investigate the efficacy of Metacognitive Training for Depression (D-MCT), a new low-threshold, modular group intervention.

DETAILED DESCRIPTION:
Despite the existence of evidence-based treatment methods, a significant treatment gap remains for major depression. While in acute psychiatric treatment of severely depressed patients a pharmacological treatment is usually applied, depression-specific psychotherapeutic (group) concepts are rarely part of the treatment, though recommended in clinical guidelines. A main reason is that present group concepts were designed primarily for outpatient settings and do not meet the structural requirements of inpatient care (i.e., short residence time, continuous admissions and dismissals).

Metacognitive Training for Depression (D-MCT) is a new low-threshold, modular group intervention which was designed to fill this treatment gap by addressing contextual and structural shortcomings of existing concepts for the use in inpatient treatment. The training targets depressive symptoms by changing (meta-) cognitive biases identified in both cognitive models of depression and basic research. D-MCT was positively evaluated with regard to feasibility and acceptance in a non-randomized pilot study.

Aim of the present randomized-controlled trial is to investigate the efficacy of D-MCT as an add-on intervention in inpatient treatment of depressed patients compared with a standard add-on group therapy (Positivity Training, PT). Based on a power analysis, the investigators target a sample size of 60 depressed patients, who will be randomized either to D-MCT or PT. Blind to diagnostic status, symptom level as well as cognitive biases will be assessed pre- and post-treatment (8 group sessions) as well as 3 months later (follow-up). Primary outcome parameter is severity of depressive symptoms measured with the HDRS total score (17-item version). Secondary outcome measures are self-assessed depression (BDI), dysfunctional beliefs (DAS), metacognitions (MCQ), self-esteem (RSE), and quality of life (WHOQOL-BREF).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depression according to DSM-IV (MINI Interview)
* Diagnosis of Dysthymia according to DSM-IV (MINI Interview)

  * DSM-IV = The Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition, Text Revision (American Psychiatric Association, 2000)

Exclusion Criteria:

* Lifetime psychotic symptoms (i.e., hallucinations, delusions, or bipolar disorder) according to DSM-IV (MINI Interview)
* Current substance dependency according to DSM-IV (MINI Interview)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HDRS), total score from pre to post treatment (4 weeks) and follow-up (3months) | 4 months
  Clinician-rated severity of depressive symptoms, 17-item version, most commonly used interview-based measure of depression

SECONDARY OUTCOMES:
Change in Beck Depression Inventory (BDI), total score from pre to post treatment (4 weeks) and follow-up (3months) | 4 months
  Self-assessed severity of depressive symptoms (questionnaire)
Change in Dysfunctional Attitudes Scale (DAS) from pre to post treatment (4 weeks) and follow-up (3months) | 4 months
  questionnaire
Change in Metacognitions Questionnaire (MCQ-30) from pre to post treatment (4 weeks) and follow-up (3months) | 4 months
  questionnaire
Change in Ruminative Responses Scale (RRS) from pre to post treatment (4 weeks) and follow-up (3months) | 4 months
  questionnaire
Change in Rosenberg Self-Esteem-Scale (RSE) from pre to post treatment (4 weeks) and follow-up (3months) | 4 months
  questionnaire
Change in quality of life (WHOQOL-BREF) from pre to post treatment (4 weeks) and follow-up (3months) | 4 months
  questionnaire
Change in coping (Brief-Cope) from pre to post treatment (4 weeks) and follow-up (3months) | 4 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marit Hauschildt, Ph.D., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Jelinek L, Otte C, Arlt, S, Hauschildt M. Denkverzerrungen erkennen und korrigieren: Eine Machbarkeitsstudie zum Metakognitiven Training bei Depressionen (D-MKT). Zeitschrift für Psychiatrie und Psychotherapie, 61(4): 1-8, 2014.